CLINICAL TRIAL: NCT02187887
Title: Brief Online Intervention to Reduce Heavy Alcohol Use Among Young Adult Veterans
Brief Title: Online Program for Young Adult Veteran Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34AA022400 (NIH); R34AA022400 (NIH)
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2019-05

CONDITIONS: AOD Misuse; AOD Associated Consequences
Keywords: alcohol; young adult veterans; brief intervention; online; perceived norms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized normative feedback (Experimental): Intervention participants receive feedback correcting their misperceptions of the drinking behavior and attitudes of fellow veterans
  Interventions: Behavioral: Personalized normative feedback
- Control (No Intervention): Control participants receive feedback correcting their misperceptions of the video game playing behavior and attitudes of fellow veterans

INTERVENTIONS:
Behavioral: Personalized normative feedback — Participants receive behavioral norms feedback based on their response to items in a baseline survey. Personal responses are presented along with perceptions of other same gender veterans and actual drinking norms of same gender veterans.
  Other Names: PNF
  Arms: Personalized normative feedback

SUMMARY:
The primary objective of the research study is to test the feasibility of a brief Internet-based intervention to reduce heavy alcohol use among young adult veterans of wars in Iraq and Afghanistan. Veterans are recruited through the social media website Facebook in two phases. In the first phase, investigators collect data from 800 veteran participants to document and analyze drinking norms in this population. In the second phase, investigators use the norms collected in Phase 1 and information from the analyses to develop and pilot test an online intervention with young adult veteran participants. Six hundred participants are recruited through Facebook and randomly assigned to intervention (N = 300) or control (N = 300) conditions. It is hypothesized that those in the intervention condition will drink less at a one-month follow-up period than those in the control condition. Investigators also collect feedback from participants on the usability of the online intervention.

DETAILED DESCRIPTION:
This study was conducted in two phases with the main goal of developing and testing a very brief online program to reduce heavy alcohol use among young adult veterans in the United States.

In the first phase, we examined how the social media website Facebook could be used to reach veterans in the community for the intervention effort. Although veterans are an at-risk group for heavy drinking and mental health problems, few seek care. Thus, we were able to document that targeted Facebook advertisements can be used to reach out to veterans and provide them with an alcohol reduction program that they likely would not have received otherwise.

In the second phase, we used the data we collected from participants in the first phase to develop a personalized normative feedback intervention. This intervention was very brief and online, and showed young veterans information to correct their misperceptions about the drinking behavior of their peers. For example, in the intervention, young veterans would be asked how much they believe other veterans like themselves drink alcohol. Then, they would view information about veterans like themselves that showed them that other veterans do not drink as much as they think they do. This is important because much research has documented that perceptions about how much others drink is a major factor contributing to how much one drinks themselves. Thus, correcting these misperceptions has been a primary strategy for reducing drinking among young people. These norms correction strategies have mostly been tested with college students or other non-veteran young adult groups, and when they have been tested with veterans they have been tested within much lengthier, multicomponent interventions. Our study was the first to test the norms correction strategy alone with young veterans using an online design meant to reach veterans in the community through recruitment on Facebook.

ELIGIBILITY:
Inclusion Criteria:

1. United States veteran from Operation Enduring Freedom, Operation Iraqi Freedom, or Operation New Dawn who has been discharged or separated from the Army, Navy, Marines, or Air Force and is not currently in the reserves
2. between the ages of 18 and 34
3. the ability to read English (also a requirement of military service)
4. access to a computer and the Internet
5. has an email address 6) an AUDIT score of >4 (men) or >3 (women) in order to reach those who may benefit from an intervention targeted toward reducing alcohol misuse

Exclusion Criteria:

* None besides not meeting inclusion criteria

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 793 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Pedersen, PhD, Principal Investigator — RAND
Locations (1):
- RAND, Santa Monica, California, United States

REFERENCES:
- [Derived] Pedersen ER, Marshall GN, Schell TL. Study protocol for a web-based personalized normative feedback alcohol intervention for young adult veterans. Addict Sci Clin Pract. 2016 Mar 31;11(1):6. doi: 10.1186/s13722-016-0055-8. PMID 27036408
- [Derived] Pedersen ER, Helmuth ED, Marshall GN, Schell TL, PunKay M, Kurz J. Using facebook to recruit young adult veterans: online mental health research. JMIR Res Protoc. 2015 Jun 1;4(2):e63. doi: 10.2196/resprot.3996. PMID 26033209

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Personalized Normative Feedback | Control
Started | 393 | 400
Completed | 388 | 396
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Normative Feedback | Control | Total
Number analyzed (Participants) | 388 | 396 | 784
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (3.3) | 28.9 (3.5) | 28.9 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 70 | 131
  Male | 327 | 326 | 653
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 46 | 82
  Not Hispanic or Latino | 352 | 350 | 702
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 10 | 19
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 14 | 18 | 32
  White | 330 | 334 | 664
  More than one race | 25 | 20 | 45
  Unknown or Not Reported | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Total drinks per week in the past 30 days
Time Frame: Past month (30 days)
Measure: Mean (Standard Deviation); unit: drinks per week at follow-up month
Arm/Group | Personalized Normative Feedback | Control
Number analyzed (Participants) | 388 | 396
drinks per week at follow-up month | 9.9 (12.1) | 13.4 (14.8)

2. Primary Outcome: Alcohol-related Consequences
Description: Brief Young Adult Alcohol Consequences Questionnaire. This is a 21 item measure of alcohol-related consequences experienced by young adults. Participants indicate whether or not they have experienced each of the consequences in the past month (1 = yes, 0 = no). Scores range from 0 to 21 with higher scores indicated a greater number of consequences experienced.
  Citation: Kahler, C. W., Strong, D. R., & Read, J. P. (2005). Toward efficient and comprehensive measurement of the alcohol problems continuum in college students: The Brief Young Adult Alcohol Consequences Questionnaire. Alcoholism: Clinical and Experimental Research, 29(7), 1180-1189.
Time Frame: Past month (30 days)
Measure: Mean (Standard Deviation); unit: consequences at follow-up month
Arm/Group | Personalized Normative Feedback | Control
Number analyzed (Participants) | 388 | 396
consequences at follow-up month | 3.8 (5.6) | 5.3 (6.3)

ADVERSE EVENTS:
Arm/Group | Personalized Normative Feedback | Control
Serious Adverse Events (participants affected / at risk) | 0/388 | 0/396
Other Adverse Events (participants affected / at risk) | 0/388 | 0/396

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No